CLINICAL TRIAL: NCT06432595
Title: Effect of Instability Resistance Training on Balance, Core Muscle Strength, and Athletic Performance Among Young Male Chinese Kayak Canoeists
Brief Title: Effect of Instability Resistance Training on Balance, Core Muscle Strength, and Athletic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Jianxin Gao, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: JKEUPM-2023-256
Record Dates: First submitted 2024-01-07; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Athletic Performance
Keywords: Instability resistance training; Balance ability; Core muscle strength; Athletic performance; Kayak canoeists

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instability resistance training (Experimental): After pre-testing, participants were randomly assigned to two groups. The participants of the IRT group were conducted in a 12-week (July 3 to September 22, 2023) Instability resistance training program that was performed one hour and three times per week (Mondays, Wednesdays, and Fridays from 4 to 5 pm) in the Nanchang Yao Lake base.
  Interventions: Other: Instability resistance training and Traditional resistance training
- Traditional resistance training (Experimental): After pre-testing, participants were randomly assigned to two groups. The participants of the TRT group were conducted in a 12-week (July 3 to September 22, 2023) traditional resistance training program that was performed one hour and three times per week (Mondays, Wednesdays, and Fridays from 4 to 5 pm) in the Ganzhou Shangyou base.
  Interventions: Other: Instability resistance training and Traditional resistance training

INTERVENTIONS:
Other: Instability resistance training and Traditional resistance training — The 20 intervention actions were divided into three levels (primary, intermediate, and advanced) for instability resistance training and traditional resistance training. Both groups performed training for 60 minutes three times a week. The Swiss ball, BOSU ball, and Wobble boards only provided an unstable surface environment for instability resistance training. The intensity/load was body weight for both training methods.

SUMMARY:
The goal of this experimental study is to examine the effect of instability resistance training (IRT) on balance ability, core muscle strength, and athletic performance of young Chinese male kayak canoeists. The main questions it aims to answer are:

Do the IRT and TRT methods have any effect on the subject's balance ability in terms of static balance and dynamic balance? Do the IRT and TRT methods have any effect on the subject's isometric strength of the core muscle group in terms of abdomen, back, left lateral, and right lateral? Do the IRT and TRT methods have any effect on the subject's isotonic strength of the core muscle group in terms of flexion, extension, left lateral flexion, and right lateral flexion? Do the IRT and TRT methods have any effect on the subject's athletic performance in terms of dynamometer performance and calm-water performance?

Researchers will compare the effect of instability resistance training (IRT) and traditional resistance training (TRT) on balance ability, core muscle strength, and athletic performance of young Chinese male kayak canoeists.

Participants will:

Take 12-week instability resistance training (IRT) and traditional resistance training (TRT) difficulty level (primary level 1-4 weeks, intermediate level 5-8 weeks, and advanced-level 9-12 weeks).

Take 3 training sessions per week and complete the training on Mondays, Wednesdays, and Fridays from 4 to 5 pm.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of a 12-week IRT on balance, core strength, and athletic performance among young male Chinese kayak canoeists. A Cluster Randomized Controlled Trial (CRCT) study was conducted. Firstly, the 2 city-level representative teams were chosen from 4 city-level representative teams of Jiangxi province and randomly assigned as two groups (experimental group and control group) using the Lottery Method. Secondly, 64 eligible kayak canoeists between the ages of 16-22 years (19.10±1.38) were recruited from the selected 2 city-level representative teams and randomly assigned to the instability resistance training (IRT) for the experimental group and traditional resistance training (TRT) for the control group using the same Lottery Method. The intervention was divided into 3 levels (primary, intermediate, and advanced) for IRT and TRT. Both groups performed training for 60 minutes, three times a week. The Swiss ball, BOSU ball, and Wobble boards were only provided with unstable surfaces for the IRT group. The intensity was body weight for both training methods. Dependent variables involving balance, core muscle strength, and athletic performance were measured using Flamingo Balance Test (FBT), Star Excursion Balance Test (SEBT), Abdomen Bridge (AB), Back Bridge (BB), Left and Right Lateral Bridge (LLB and RLB), 1min Sit-Up (SU), 1min Back Hyperextension (BH), 1min Left and Right Lateral V-up (LLV and RLV), K-1 200m Dynamometer Performance (DP), and Men's K-1 200m Calm-Water Performance (CWP) tests respectively in pre-test, post-test 1 (week 6), post-test 2 (week 12).

ELIGIBILITY:
Inclusion Criteria:

Male, Aged 16-22, and Healthy

Exclusion Criteria:

Athletes who are systematically training their balance ability and core muscle strength

Ages: 16 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Static Balance | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Flamingo Balance Test
Dynamic Balance | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Star Excursion Balance Test
Abdomen Core Strength | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Abdomen Bridge
Back Core Strength | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Back Bridge
Left Lateral Core Strength | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Left Lateral Bridge
Right Lateral Core Strength | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Right Lateral Bridge
Dynamometer Performance | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Men's K-1 200m Dynamometer Performance
Calm-Water Performance | This study collected data in pre-test (before intervention), post-test 1 (6 weeks after intervention), and post-test 2 (12 weeks after intervention)
  Men's K-1 200m Calm-Water Performance

CONTACTS AND LOCATIONS:
Locations (1):
- Jianxin Gao, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao J, Gong Z, Samsudin S, Abdullah BB, Dev Omar Dev R. The effects of instability core training on balance ability and paddling performance among young male Chinese flatwater sprint kayakers: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Jul 10;17(1):191. doi: 10.1186/s13102-025-01248-6. PMID 40640954